CLINICAL TRIAL: NCT00167960
Title: Effects on the Emergence and Transmission of Vancomycin-Resistant Enterococci After Changes in Antibiotic Use in a Hematology Unit.
Brief Title: Study Evaluating Vancomycin-Resistant Enterococci in a Hematology Unit
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0910X-101525
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Gram-Positive Bacterial Infections
Keywords: Bacterial Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Bacterial Infections | interventions — Piperacillin; Tazobactam

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Drug: Piperacillin/tazobactam and other β-lactam/β-lactamase

SUMMARY:
To determine the impact of the restriction of the third and forth generation cephalosporins on the reduction of intestinal colonization or infection with vancomycin-resistant enterococci (VRE) in a surgical intensive care unit (SICU)

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to or transferred to the SICU.
* Eligible patients will be patients of either sex, 18 years of age or older who are admitted or transferred to the SICU.
* Provide written informed consent

Exclusion Criteria:

* Patients who have hypersensitivity to penicillin, cephalosporins or beta-lactamase inhibitors.
* Females who are pregnant and breast feeding
* Any underlying conditions or non-infectious diseases that will be ultimately fatal within 48 hours.
* Those who have already been participating other clinical study related with antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- South Korea (2):
  - Incheon
  - Ulsan